CLINICAL TRIAL: NCT01538030
Title: Perinatal Outcomes According to Amniotic Fluid Indez After Premature Rupture of Membranes. A Prospective Cohort Study.
Brief Title: Perinatal Outcome After Premature Rupture of Membranes
Status: Completed | Type: Observational
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Other Study IDs: MHST2012-03
Record Dates: First submitted 2012-02-18; First posted 2012-02-23 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Fetal Membranes; Premature Rupture
Keywords: Fetal membranes, premature rupture; Cesarean section; Perinatal mortality; Neonatal sepsis; Amniotic Fluid Volume
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Perinatal Death; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amniotic Fluid Volume > 5: Pregnant patients with gestations between 24-34 weeks with premature rupture of membranes that, when the decision was made to interrupt the pregnancy, had amniotic fluid volume index above 5.1
- Amniotic Fluid Volume < 5: Pregnant patients with gestations between 24-34 weeks with premature rupture of membranes that, when the decision was made to interrupt the pregnancy, had amniotic fluid volume index of 5 or less.

SUMMARY:
Premature rupture of membranes is an important cause of neonatal morbidity and mortality, mainly because of the complications associated with this pathology (oligohydramnios, cord compression or prolapse, infection). When rupture of the membranes occur the risk of cord compression increases but there is little evidence regarding this complication and amniotic fluid volume. The investigator's focus are the perinatal outcomes according to amniotic fluid volume (< 5 or >5).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24-34 weeks.
* Confirmed diagnosis of premature rupture of membranes.

Exclusion Criteria:

* Twin pregnancies.
* Obstetric pathologies that require immediate termination of pregnancy (severe preeclampsia, abruptio placenta, cord prolapse).
* Termination of pregnancy (whatever the reason) before complete corticoid treatment.
* Incomplete recollection of all data required for analysis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients between 24-34 weeks of gestation with a confirmed diagnosis of premature rupture of membranes.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cesarean section rate | 5 months
  Number of cases in each cohort that were interrupted by cesarean section due to fetal distress (evidence of cord dystocia).

SECONDARY OUTCOMES:
Perinatal mortality | 5 months
  Number of perinatal deaths (ante, peri and postpartum until 28 days postpartum)in each cohort.
Neonatal sepsis | 5 months
  Number of cases of neonates diagnosed with sepsis in each cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama